CLINICAL TRIAL: NCT03696719
Title: Anesthetic Method and Cerebral Outcomes: A Prospective Randomized Controlled Trial.
Brief Title: Anesthetic Method and Cerebral Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Leonid Eidelman, Professor, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 616-18
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia; Neuron Degeneration
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Undergoing surgery under general anesthesia (Active Comparator): Patients will undergo the surgery under general anesthesia, anesthetic regime will be according to standard clinical practice.
  Interventions: Device: BIS bispectral index monitoring device; Biological: NSE cerebral biomarker testing
- Undergoing surgery under regional anesthesia (Active Comparator): Patients will undergo the surgery under neuroaxial anesthesia.
  Interventions: Biological: NSE cerebral biomarker testing

INTERVENTIONS:
Device: BIS bispectral index monitoring device — In addition to the standard monitoring prescribed by the American society of Anesthesiologists, all study participants will be monitored with the BIS, a noninvasive monitoring device which measures the depth of anesthesia. The monitoring is performed using noninvasive electrodes placed on the forehead.
  Arms: Undergoing surgery under general anesthesia
Biological: NSE cerebral biomarker testing — Venous blood will be collected from each participant in the surgery room prior to anesthesia induction, throughout anesthesia and one hour following surgery in the PACU in order to assess NSE cerebral biomarker according to the ELISA method requirements. At each one of the assessment points 9 cc of venous of blood will be taken from each of the study participants, while routine blood tests are taken.

SUMMARY:
Research regarding the effects of anesthesia on the central nervous system remain controversial with some studies suggesting a neurotoxic effect and others indicating a neuroprotective effect.

In recent years numerous neuronal proteins have been found to be useful tools for diagnosis and prognosis of cerebral tissue damage. Among these neuronal proteins are the following markers: Neuron Specific Enolase (NSE), Tau protein, Glial Fibrillary Acidic Protein (GFAP), Ubiquitin Carboxy-Hydrolase L1 (UCH-L1).

BIS is a non-invasive brain monitoring technology which monitors the depth of anesthesia.

In this randomized clinical trial, we aim to examine the effect of anesthetic method (General anesthesia and neuroaxial anesthesia) on neuronal damage as measured by NSE serum levels.

One hundred and forty patients aged 18 and above undergoing Transurethral resection of the prostate, Trans Urethral Resection of the Bladder Tumor, Tension Free Vaginal Tap , Trans Obturator Tension Free Vaginal Tap and pelvic floor repair surgeries will be enrolled in the study.

Patients will randomly be assigned to undergo the study either under general anesthesia or with neuroaxial anesthesia.

Participants will be monitored using the BIS monitor, to measure the depth of anesthesia.

Additionally, 9 cc of venous blood be collected from each participant in the surgery room prior to anesthesia induction, throughout anesthesia and one hour following surgery in the PACU in order to assess NSE levels.

DETAILED DESCRIPTION:
I

Specific Aim:

Primary Endpoint Our primary endpoint is to compare the effect of anesthetic method (GA vs. NA) on plasma level of neuronal damage biomarker NSE.

Study Design:

This is a prospective, single center, randomized controlled trial that try to assess the effect of anesthetic method on neuronal damage biomarker level. The study will be conducted at the Rabin Medical Center (Beilinson Campus), Petach Tikva, Israel, a tertiary university hospital.

One hundred and forty patients aged 18 and above, undergoing elective TURB, TURBT, (TVT-O) and pelvic floor repair surgeries, will be enrolled in the study following providing their consent for participation.

Index procedure:

After consenting to participation patients will be randomly assigned to one of the following study groups:

1. Patients undergoing surgery under GA
2. Patients undergoing surgery with NA. Anesthetic regime will be subject to standard clinical guidelines and to clinical judgement of the attending anesthesiologist.

Intraoperative and postoperative hemodynamic monitoring will be according to standard departmental and clinical guidelines. Data will be recorded and stored electronically by Metavision system (iMDsoft company).

BIS monitoring:

In addition to the standard monitoring prescribed by the American society of Anesthesiologists, all study participants will be monitored with the BIS, a noninvasive monitoring device which measures the depth of anesthesia. The monitoring is performed using noninvasive electrodes placed on the forehead.

Blood tests:

Venous blood will be collected from each participant in the surgery room prior to anesthesia induction, throughout anesthesia and one hour following surgery in the PACU in order to assess cerebral biomarkers according to the ELISA method requirements. At each one of the assessment points 9 cc of venous of blood will be taken from each of the study participants, while routine blood tests are taken.

Data Collection

For each participating patient the following data will be collected and recorded through the study duration:

1. Demographic data
2. Each participant medical history including concomitant medications.
3. Hemodynamic data including heart rate, automatic non-invasive blood pressure measurements, temperature as well pulse oximetry as routine procedures will be recorded and stored by Metavision system.
4. Anesthetic data: anesthetic method, anesthetic agents given throughout surgery, anesthetic complications.
5. Opioid use in the first 24 hours after surgery.
6. Duration of stay in the PACU.
7. Duration of hospital stay
8. Functional status upon hospital release.

ELIGIBILITY:
Inclusion Criteria:

The study will conducted in Beilinson Hospital . All patients above 18 presenting for primary TURP, TURBT, TVT, TVT-O and pelvic floor repair surgeries. All patients who are able to comply with the study requirements and gave a written informed consents.

Exclusion Criteria:

1. Patients with a history of a cerebrovascular accident (CVA) or Transient ischemic attack (TIA) in the year prior to surgery.
2. Patients with significant decreases in cognitive function prior to surgery.
3. Patients presenting for a secondary TURB surgery.
4. Patient with a contraindication to NA.
5. Patients who are unable to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
NSE serum level in PACU | 1 hour after surgery completion

SECONDARY OUTCOMES:
NSE serum levels after anesthesia induction | Half an hour after anesthesia induction

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center/Beilinson Campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Evered L, Silbert B, Scott DA, Zetterberg H, Blennow K. Association of Changes in Plasma Neurofilament Light and Tau Levels With Anesthesia and Surgery: Results From the CAPACITY and ARCADIAN Studies. JAMA Neurol. 2018 May 1;75(5):542-547. doi: 10.1001/jamaneurol.2017.4913. PMID 29459944
- [Background] Cata JP, Abdelmalak B, Farag E. Neurological biomarkers in the perioperative period. Br J Anaesth. 2011 Dec;107(6):844-58. doi: 10.1093/bja/aer338. Epub 2011 Nov 6. PMID 22065690
- [Background] Tomaszewski D. Biomarkers of Brain Damage and Postoperative Cognitive Disorders in Orthopedic Patients: An Update. Biomed Res Int. 2015;2015:402959. doi: 10.1155/2015/402959. Epub 2015 Aug 31. PMID 26417595
- [Background] Trakas E, Domnina Y, Panigrahy A, Baust T, Callahan PM, Morell VO, Munoz R, Bell MJ, Sanchez-de-Toledo J. Serum Neuronal Biomarkers in Neonates With Congenital Heart Disease Undergoing Cardiac Surgery. Pediatr Neurol. 2017 Jul;72:56-61. doi: 10.1016/j.pediatrneurol.2017.04.011. Epub 2017 Apr 21. PMID 28571730
- [Background] van Munster BC, Korse CM, de Rooij SE, Bonfrer JM, Zwinderman AH, Korevaar JC. Markers of cerebral damage during delirium in elderly patients with hip fracture. BMC Neurol. 2009 May 27;9:21. doi: 10.1186/1471-2377-9-21. PMID 19473521
- [Background] Rappold T, Laflam A, Hori D, Brown C, Brandt J, Mintz CD, Sieber F, Gottschalk A, Yenokyan G, Everett A, Hogue CW. Evidence of an association between brain cellular injury and cognitive decline after non-cardiac surgery. Br J Anaesth. 2016 Jan;116(1):83-9. doi: 10.1093/bja/aev415. PMID 26675953
- [Background] Li YN, Zhang Q, Yin CP, Guo YY, Huo SP, Wang L, Wang QJ. Effects of nimodipine on postoperative delirium in elderly under general anesthesia: A prospective, randomized, controlled clinical trial. Medicine (Baltimore). 2017 May;96(19):e6849. doi: 10.1097/MD.0000000000006849. PMID 28489775
- [Background] Yokobori S, Hosein K, Burks S, Sharma I, Gajavelli S, Bullock R. Biomarkers for the clinical differential diagnosis in traumatic brain injury--a systematic review. CNS Neurosci Ther. 2013 Aug;19(8):556-65. doi: 10.1111/cns.12127. Epub 2013 May 27. PMID 23710877
- [Background] Feng F, Chen Z, Cromer J, Doerr A, Glow A, Horstman-Reser A, Infanger A, Lovas E, Ryberg J, Sinclair M, Zecy A. Anesthetic Concerns for Patients Undergoing a Transurethral Resection of the Prostate (TURP). Urol Nurs. 2016 Mar-Apr;36(2):75-81. PMID 27281864
- [Background] Jang D, Lim CS, Shin YS, Ko YK, Park SI, Song SH, Kim BJ. A comparison of regional and general anesthesia effects on 5 year survival and cancer recurrence after transurethral resection of the bladder tumor: a retrospective analysis. BMC Anesthesiol. 2016 Mar 12;16:16. doi: 10.1186/s12871-016-0181-6. PMID 26971194
- [Background] Ballard C, Jones E, Gauge N, Aarsland D, Nilsen OB, Saxby BK, Lowery D, Corbett A, Wesnes K, Katsaiti E, Arden J, Amoako D, Prophet N, Purushothaman B, Green D. Optimised anaesthesia to reduce post operative cognitive decline (POCD) in older patients undergoing elective surgery, a randomised controlled trial. PLoS One. 2012;7(6):e37410. doi: 10.1371/journal.pone.0037410. Epub 2012 Jun 15. PMID 22719840